CLINICAL TRIAL: NCT03303742
Title: Evaluation of Patient Satisfaction, Color Difference, Marginal Integrity and Survival of Bruxzir Zirconia Complete Coverage Crowns With Feather Edge Versus Deep Chamfer Finish Line Marginal Design.
Brief Title: Feather Edge Versus Deep Chamfer Finish Line Marginal Design in Complete Coverage Bruxzir Zirconia Crowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Elbasha, assistant lecturer of fixed prosthodontics/ahram canadian university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-10-03
Record Dates: First submitted 2017-10-03; First posted 2017-10-06 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Premolars Need Full Coverage Restoration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- feather edge finish line marginal design (Experimental): intervention
  Interventions: Other: feather edge
- deep chamfer finish line marginal design (Active Comparator): comparator
  Interventions: Other: deep chamfer

INTERVENTIONS:
Other: deep chamfer — finish line marginal design of a full coverage crown preparation
  Other Names: rounded shoulder
  Arms: deep chamfer finish line marginal design
Other: feather edge — finish line marginal design of a full coverage crown preparation
  Other Names: knife edge
  Arms: feather edge finish line marginal design

SUMMARY:
Evaluation of patient satisfaction, color difference, marginal integrity and survival of Bruxzir Zirconia complete coverage crowns with feather edge versus deep chamfer finish line marginal design.

(Randomised Controlled Trial)

ELIGIBILITY:
Inclusion Criteria:

* 19-50 years.
* Males or females.
* Co-operative patients approving to participate in the trial.

Exclusion Criteria:

* Patients younger than 19 years old
* Disabilities
* Systemic diseases or severe medically compromised
* Lack of compliance of the patient contributed in the study

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-08-10 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | one year
  patient satisfaction will be measured by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Sara Hussein Elbasha, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided